CLINICAL TRIAL: NCT02591511
Title: Effects of Health-education Application on Improving Stroke-related Knowledge and Health Related Quality of Life in Patients With Stroke: a Randomized Controlled Trial
Brief Title: Effects of Patient-centered Stroke Educating System: a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Taipei Medical University
Record Dates: First submitted 2015-10-28; First posted 2015-10-29 (Estimated); Results first posted 2018-09-14 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2015-10

CONDITIONS: Health Education
MeSH Terms: conditions — Health Education

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- health-education app (Experimental): Smart phone and pad is a stroke-related health education app intervention group
  Interventions: Device: smart phone and pad
- health education manuals (Active Comparator): stroke-related health education manual control group
  Interventions: Other: stroke-related health education manual

INTERVENTIONS:
Device: smart phone and pad — Smart phone and pad is the mobile include the smart phone and pad, that can download the APP from internet.
  Arms: health-education app
Other: stroke-related health education manual — stroke-related health education manual is the manual mainly contained information regarding the prevention of stroke risk factors.
  Arms: health education manuals

SUMMARY:
The aim of this study is to establish PAtient-Centered Computerized Educating System for Stroke (PACCESS) for patients with different demands and lack of knowledge.Those in the intervention group will receive the PACCESS and the control groups will receive traditional health education to test the effects of PACCESS in increasing clinical decision-making, health behavior, activities of daily living and knowledge of stroke, and health care quality.

DETAILED DESCRIPTION:
To prevent recurrent stroke and improve the health-related quality of life (HRQOL) in patients with stroke, education regarding the risk factors of recurrent stroke is a crucial part of effective care for patients with stroke. The aim of this study was to develop an application capable of providing health education for recurrent-stroke prevention. We also examined the effectiveness of this app for improving stroke-related knowledge and HRQOL in patients with stroke.

ELIGIBILITY:
Inclusion Criteria:

* first time diagnosis of stroke (International Classification of Diseases, ninth revision, clinical modification [ICD-9] codes) of cerebral hemorrhage (ICD-9, 431) or cerebral infarction (ICD 9, 434)
* ability to follow instructions and complete the interviews
* having a designated caregiver who agrees to participate in the survey
* >6 years of education
* have smartphone or the other mobile device can download the APP from internet.

Exclusion Criteria:

* cognitive impairment (Mini-Mental State Examination (MMSE scores<24)
* having major mental diseases (i.e., depression, dementia, delirium, etc.)
* the inability to read/answer questionnaires

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Hsuan Hou, PHD, Study Chair — Taipei Medical University

REFERENCES:
- [Derived] Crocker TF, Brown L, Lam N, Wray F, Knapp P, Forster A. Information provision for stroke survivors and their carers. Cochrane Database Syst Rev. 2021 Nov 23;11(11):CD001919. doi: 10.1002/14651858.CD001919.pub4. PMID 34813082
- [Derived] Kang YN, Shen HN, Lin CY, Elwyn G, Huang SC, Wu TF, Hou WH. Does a Mobile app improve patients' knowledge of stroke risk factors and health-related quality of life in patients with stroke? A randomized controlled trial. BMC Med Inform Decis Mak. 2019 Dec 21;19(1):282. doi: 10.1186/s12911-019-1000-z. PMID 31864348

RESULTS

PARTICIPANT FLOW:
Groups:
- Health-education App: 1. assisting the subjects in installing the app onto their personal smartphones;
  2. teaching the patients about the content of the app and explaining its method of operation
- Health Education Manuals: 1. giving the stroke-related health education manuals to subjects;
  2. teaching the patients about the content of the manual.
Period: Overall Study
Arm/Group | Health-education App | Health Education Manuals
Started | 30 | 33
Completed | 30 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Health-education App: (1) assisting the subjects in installing the app onto their personal smartphones; (2) teaching the patients about the content of the app and explaining its method of operation.
- Health Education Manuals: (1) giving the stroke-related health education manuals to subjects; (2) teaching the patients about the content of the manual.
- Total: Total of all reporting groups
Arm/Group | Health-education App | Health Education Manuals | Total
Number analyzed (Participants) | 30 | 33 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 23 | 43
  >=65 years | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.47 (10.82) | 52.33 (11.33) | 51.40 (11.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 21 | 22 | 43
Region of Enrollment [Number; unit: participants]
  Taiwan | 30 | 33 | 63
Stroke knowledge questionnaire [Mean (Standard Deviation); unit: participants] | 26.23 (6.65) | 25.21 (5.54) | 25.72 (6.10)

OUTCOME MEASURES:

1. Primary Outcome: Stroke Health Education Knowledge Questionnaire
Description: The stroke knowledge questionnaire is the primary outcome of this study. The questions are single-choice questions. The content of the questions are based on the stroke health education manual and adapted to APP format in this study. For the 12 risk factors, each risk factor was sorted out 3 questions. There are total of 36 (3x12 = 36) questions of stroke knowledge, a score of 1 for each question, the highest score of 3 for each risk factor, the highest score of 36 points and the lowest score of 0 point. The higher score represents the better outcome.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Health-education App | Health Education Manuals
Number analyzed (Participants) | 30 | 33
score on a scale | 29.07 (5.27) | 28.00 (5.46)

ADVERSE EVENTS:
Time Frame: 3 months
Groups:
- Health Education Manual: (1) giving the stroke-related health education manuals to subjects; (2) teaching the patients about the content of the manual.
Arm/Group | Health-education App | Health Education Manual
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/33
Other Adverse Events (participants affected / at risk) | 0/30 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less